CLINICAL TRIAL: NCT00637611
Title: Single-Center, Double-Blind, Randomized , Parallel Study Comparing Onset of Action, Efficacy & Safety of a Single-Dose of Fexofenadine HCl 180 mg vs Montelukast Na 10 mg & Placebo in Treating Seasonal Allergic Rhinitis Subjects in an Allergen Exposure Unit (Study I)
Brief Title: Single-Center, Double-Blind, Randomized , Parallel Study Comparing Onset of Action, Efficacy & Safety of a Single-Dose of Fexofenadine HCl 180 mg vs Montelukast Na 10 mg & Placebo in Treating Seasonal Allergic Rhinitis Subjects in an Allergen Exposure Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A_4149
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine HCl
  Other Names: Allegra

SUMMARY:
The primary objective of this study is to determine the efficacy and onsets of action of single-dose fexofenadine hydrochloride 180 mg and montelukast sodium 10 mg relative to placebo. Secondary objectives are to compare the safety and efficacy of fexofenadine hydrochloride 180 mg, montelukast sodium 10 mg, and placebo

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 15 years of age or older
* History of seasonal allergic rhinitis (SAR) during the fall pollen season, for at least the previous 2 years
* History of having a positive response to antihistamines for symptoms of SAR
* Must be skin test positive to ragweed within the last 15 months with at least a moderate reaction as defined by a wheal 7 mm greater than the diluent wheal after intradermal skin test or a wheal 5 mm greater than the diluent wheal after skin prick test. A skin test performed in the previous 15 months may be used to qualify the patient if it was performed at the investigator's site and recorded in the subject's medical record
* All females must have negative urine pregnancy test at screening visit
* Willing and able to adhere to visit schedules and all study requirements

Exclusion Criteria:

* Clinically significant medical condition (such as cardiovascular, hepatic, neurologic, hematological, renal, gastrointestinal, endocrine, or other major systemic disease), which, in the judgment of the investigator, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult
* Asthma that requires treatment with medication other than an inhaled, short-acting beta agonist or asthma that will be exacerbated by exposure to ragweed pollen
* Pregnancy or breast-feeding
* History of hypersensitivity to the study medications or to drugs with similar chemical structures
* Nasal structural abnormalities, including large nasal polyps or marked septal deviation, that significantly interfere with nasal air flow
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Upper or lower respiratory infection within 14 days of the first priming visit
* Diagnosis of sinusitis within 30 days of the first priming visit
* Immunotherapy, except those on a constant dose of immunotherapy that will be maintained throughout the study
* Treatment with any investigational drug in the last 30 days before study entry
* Recent history of drug or alcohol abuse
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Unlikelihood to comply with protocol such as those with uncooperative attitude or the inability to return for follow-up visits or to complete the study
* Subjects who were randomized into this trial will not be eligible to participate in another fexofenadine hydrochloride 180 mg vs montelukast sodium 10 mg onset of action study (planned to be conducted in 2003)
* Subjects who are research employees or relatives of study site staff involved in this study or those who have or will read the protocol

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2003-02; Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy and onsets of action of single-dose fexofenadine hydrochloride 180 mg and montelukast sodium 10 mg relative to placebo in the treatment of subjects with moderately severe seasonal allergic rhinitis (SAR) in a controlled setting.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States